CLINICAL TRIAL: NCT01255826
Title: Ventilatory Management of the Preterm Neonate in the Delivery Room.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Mohamed Mohamed Shinkar, MD, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Dina Shinkar MD protocol; Sustianed inflation trial (Registry Identifier: Sustianed inflation trial)
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: Preterm; Neonates; Delivery room; Resuscitation; Ventilation; Neopuff; CPAP
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sustained lung inflation followed by CPAP (Active Comparator): Sustained pressure-controlled inflation using a neonatal mask and a T-piece ventilator (NeoPuff Infant Resuscitator; Fisher & Paykel, Auckland, New Zealand).
  This will be followed by early CPAP.
  Interventions: Procedure: Resuscitation of preterm neonates by sustained lung inflation through T piece device followed by CPAP
- Conventional self inflating bag and mask ventilation (Active Comparator): Intermittent bag and mask ventilation using a self-inflating bag with an oxygen reservoir.
  Interventions: Procedure: Resuscitation of preterm neonates by intermittent bag and mask ventilation using self inflating bag.

INTERVENTIONS:
Procedure: Resuscitation of preterm neonates by sustained lung inflation through T piece device followed by CPAP — After oropharyngeal and nasal suctioning, if there are no signs of spontaneous breathing or breathing is insufficient and/or heart rate is below 100 bpm, the following approach will be followed:Pressure-controlled (20 cm H2O) inflation will be sustained for 15 secs, using a neonatal mask and a T-piece ventilator (NeoPuff Infant Resuscitator; Fisher & Paykel).To avoid pressure leakage, we will use a neonatal mask of appropriate size which adequately cover both the mouth and nostrils of infants. This pressure controlled inflation will be followed by CPAP at 5 Cm H2O.This procedure will be repeated a second time with a pressure of 25 cm H2O for 15 secs if breathing remained insufficient and/or the heart rate is < 100 bpm and/or the infant is cyanotic. To be followed by CPAP at 6 Cm H2O.A third puff with a pressure of 30 cm H2O for 15 secs will be used after few seconds if inadequate heart rate and respiration was not reached. This will be followed by CPAP at 7 Cm H2O.
  Arms: Sustained lung inflation followed by CPAP
Procedure: Resuscitation of preterm neonates by intermittent bag and mask ventilation using self inflating bag. — After oropharyngeal and nasal suctioning, if there is no signs of spontaneous breathing or breathing is insufficient and/or heart rate is below 100 bpm, intermittent mask and bag ventilation will be administrated at a rate 40-60 per minute using a self-inflating bag and mask with an oxygen reservoir.
  Arms: Conventional self inflating bag and mask ventilation

SUMMARY:
The purpose of this study is to evaluate sustained lung inflation followed by early nCPAP as delivery room ventilatory management for preterm neonates at risk of respiratory distress syndrome in reducing their need for mechanical ventilation and ameliorating lung injury without inducing adverse effects compared with intermittent bag and mask ventilation.

DETAILED DESCRIPTION:
Neonatal resuscitation provides lifesaving intervention that, if properly conducted, not only can reduce mortality but probably can significantly decrease subsequent morbidity.

Premature infants need appropriate respiratory support and a lung-protective strategy, starting from the delivery room where, on the contrary, an inadequate respiratory approach may influence pulmonary outcome.

Mechanical ventilation in the form of positive pressure ventilation has remained the mainstay of treatment of respiratory distress syndrome (RDS) in preterm babies. In recent years, a number of new ventilation strategies have been introduced but the problem of bronchopulmonary dysplasia (BPD) has not been solved.

Sustained lung inflation (SLI) lead to a large increase in the tidal volume and the functional residual capacity(FCR) as this intervention may influence the clearance of lung fluids and allow a more even distribution of air throughout the lungs, thus facilitating the formation of FRC.

Nasal CPAP and early PEEP act through stabilization and subsequent recruitment of collapsed alveoli, increased FRC resulting in increased alveolar surface area for gas exchange and a decrease in intrapulmonary shunt .also it conserves endogenous surfactant.

Previous studies with promising results showed that a combination of sustained lung inflation and early nasal CPAP may be the most effective and least injurious way to recruit the lung in preterm neonates at birth.

This study will evaluate sustained lung inflation followed by early nCPAP as delivery room ventilatory management for preterm neonates at risk of respiratory distress syndrome in reducing their need for mechanical ventilation and ameliorating lung injury without inducing adverse effects compared with intermittent bag and mask ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants (gestational age < 34 weeks)

Exclusion Criteria:

* 1. Neonates with major congenital anomalies (congenital heart disease, neural tube defect, trisomy, etc.).

  2.Meconium aspiration syndrome, congenital diaphragmatic hernia and anterior abdominal wall defect.

  3.Maternal chorioamnionitis. 4.Neonates with gestational age < 26 weeks and /or birth weight less than 750 grams.

Ages: 27 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Proportionate of neonates in each group who will need endotracheal intubation after failure of positive pressure ventilation through face mask in the delivery room. | 2 minutes
Need for mechanical ventilation for neonates on nCPAP | 28 days

SECONDARY OUTCOMES:
Occurrence and duration of oxygen therapy. | 28 days
Bronchopulmonary dysplasia (BPD): defined as oxygen requirements more than 28 days. | 28 days
Pulmonary air leaks | 28 days
Patent ductus arteriosus (PDA). | 7 days
Necrotizing enterocolitis (NEC). | 28 days
Intraventricular hemorrhage (IVH). | 28 days
Neonatal sepsis. | 28 days
Length of NICU stay. | 28 days
Delivery room death or death during admission. | 28 days
Inflammatory mediators before and after resuscitation | 2 hours
  Serum Interleukin-1β (IL-1β) and Tumor Necrosis Factor-α (TNF-α)will be measured both initial cord blood before any resuscitation is done and a second time two hours after resuscitation.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Sami El Shimi, MD, Principal Investigator — Ain Shams University; Hesham Abdel Samie Awad, MD, Principal Investigator — Ain Shams University; Tarek Mohey El Gammacy, MD, Principal Investigator — Ain Shams University; Ola Galal Badr El Deen, MD, Principal Investigator — Ain Shams University; Dina Mohamed Mohamed Shinkar, MSc, Principal Investigator — Ain Shams University
Locations (1):
- Gynecology and Obstetrics hospital, Ain-Shams University, Cairo, Egypt